CLINICAL TRIAL: NCT02770378
Title: A Proof-of-concept Clinical Trial Assessing the Safety of the Coordinated Undermining of Survival Paths by 9 Repurposed Drugs Combined With Metronomic Temozolomide (CUSP9v3 Treatment Protocol) for Recurrent Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: Reliable Cancer Therapies (Industry); Anticancer Fund, Belgium (Other)
Responsible Party: Principal Investigator, Marc-Eric Halatsch, Prof. Dr., University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUSP9v3
Record Dates: First submitted 2016-03-14; First posted 2016-05-12 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Glioblastoma
Keywords: Temozolomide; Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Aprepitant; Minocycline; Disulfiram; Celecoxib; Sertraline; Captopril; Itraconazole; Ritonavir; Auranofin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temozolomide combined with 9 repurposed drugs (Experimental): After enrollment, the subject goes into the induction cycle, which lasts 35 days. The induction cycle consists of a drug-by-drug addition and up-dosing process.
  Hereafter, the subject will enter the treatment cycles (up to 12). During the induction cycle and the first 2 treatment cycles, regimen adjustments (dropping of certain drugs, dose modification of certain drugs) may be executed to accommodate to the patients' individual toxicity reactions that may occur during this period.
  Interventions: Drug: Temozolomide; Drug: Aprepitant; Drug: Minocycline; Drug: Disulfiram; Drug: Celecoxib; Drug: Sertraline; Drug: Captopril; Drug: Itraconazole; Drug: Ritonavir; Drug: Auranofin

INTERVENTIONS:
Drug: Temozolomide — Patients will receive temozolomide at a dose of 20 mg/m² BSA twice daily with start day 1 during induction and treatment cycles
Drug: Aprepitant — Patients will receive aprepitant at a dose of 80 mg p.o. once daily with start day 1 during induction and treatment cycles
Drug: Minocycline — Induction cycle day 3-4: minocycline 50 mg p.o. twice daily from day 19-20; minocycline 100 mg p.o. twice daily during treatment cycle 1-12 (28 days); minocycline 100 mg p.o. twice daily
Drug: Disulfiram — Induction cycle day 5-6: disulfiram 250 mg p.o. once daily from day 21-22; disulfiram 250 mg p.o. twice daily during treatment cycle 1-12 (28 days); disulfiram 250 mg p.o. twice daily
Drug: Celecoxib — Induction cycle day 1-35: day 7-8: celecoxib 200 mg p.o. twice daily from day 23-24; celecoxib 400 mg p.o. twice daily during treatment cycle 1-12 (28 days); celecoxib 400 mg p.o.twice daily
Drug: Sertraline — Induction cycle day 1-35: day 9-10: sertraline 50 mg p.o. twice daily, day 31-32: sertraline 100 mg p.o. twice daily; treatment cycle 1-12: sertraline 100 mg p.o. twice daily
Drug: Captopril — Induction cycle day 1-35: day 11-12: captopril 25 mg p.o. twice daily, day 25-26: captopril 50 mg p.o. twice daily; treatment cycle 1-12 (28 days): captopril 50 mg p.o. twice daily
Drug: Itraconazole — Induction cycle day 1-35: day 13-14: itraconazole 200 mg p.o. once daily day 27-28; itraconazole 200 mg p.o. twice daily; treatment cycle 1-12 (28 days): itraconazole 200 mg p.o.twice daily
Drug: Ritonavir — Induction cycle day 1-35: day 15-16: ritonavir 200 mg p.o. once daily, day 29-30: ritonavir 200 mg p.o. twice daily, day 35: ritonavir 400 mg p.o. twice daily; treatment cycle 1-12 (28 days): ritonavir 400 mg p.o. twice daily
Drug: Auranofin — Induction cycle day 1-35: day 17-18: auranofin 3 mg p.o. once daily, day 33-34 auranofin 3 mg p.o. twice daily; treatment cycle 1-12 auranofin 3 mg p.o. twice daily

SUMMARY:
A proof-of-concept clinical trial assessing the safety of the coordinated undermining of survival paths by 9 repurposed drugs combined with metronomic temozolomide (CUSP9v3 treatment protocol) for recurrent glioblastoma

DETAILED DESCRIPTION:
A proof-of-concept clinical trial assessing the safety of the coordinated undermining of survival paths by 9 repurposed drugs (aprepitant, auranofin, captopril, celecoxib, disulfiram, itraconazole, minocycline, ritonavir and sertraline) combined with metronomic temozolomide (CUSP9v3 treatment protocol) for recurrent glioblastoma. This is a phase I study for subjects of 18 years and older with glioblastoma that has relapsed after radiation and chemotherapy, as confirmed by histology and MRI.

A total of 10 patients will be treated with the CUSP9v3 treatment protocol. This is a monocentric trial: all patients will be treated at Ulm University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of glioblastoma World Health Organization (WHO) grade IV (histologically confirmed by a pathologist). Patients with prior low-grade glioma are eligible if histological transformation to WHO grade IV glioblastoma was confirmed.
* Progression (according to RANO criteria) after prior radiation and temozolomide treatment
* No more than 3 prior episodes of tumor progression
* ≥ 4 weeks between surgical resection or chemotherapy
* ≥ 12 weeks since last radiotherapy
* Patients > 18 years of age.
* Karnofsky performance status (KPS) of ≥ 70%
* Stable steroid dose for ≥ 1 week
* Hemoglobin ≥ 10 g/l
* Absolute neutrophil count (ANC) > 10³ cells/µl
* Platelet count > 100/µl
* Maximum 5 years since last Pneumovax (or equivalent) and varicella vaccination
* Serum creatinine, aspartat-aminotransferase (AST) and bilirubin ≤ 1.5 times the upper limit of normal (ULN)
* Female patients of childbearing potential with a negative pregnancy test within 7 days of initiation of study treatment. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Male and female patients of reproductive potential who agree to employ an effective method of birth control throughout the study and for up to 6 months following discontinuation of study drug. Patients must be counseled on the possibility of cryopreservation of oocytes or sperm.
* Signed informed consent prior to initiation of any study procedure (must understand, voluntarily sign the informed consent form and be able to adhere to the study visit schedule and other protocol requirements).

Exclusion Criteria:

* Female patients who are pregnant or breast-feeding
* Any uncontrolled/unstable medical condition except glioblastoma, including but not limited to uncontrolled/unstable hypertension, uncontrolled/unstable diabetes, uncontrolled endocrinopathies of any kind, uncontrolled/unstable psychiatric conditions
* Renal failure (eGFR < 60 ml/min)
* Active infection, including pneumonia as shown on X-ray
* Therapeutic anticoagulation use
* Prior stereotactic radiosurgery
* Radiation implants
* Radiolabeled monoclonal antibody therapy unless there was unequivocal disease progression (e.g. a new lesion or biopsy-confirmed recurrence)
* QT interval (QTc) < 470 msec (based on the mean value of triplicate ECGs), family or personal history of long or short QT syndrome, Brugada syndrome, or known history of QTc prolongation or Torsade de Pointes
* Uncontrolled electrolyte disorders that can aggravate the effects of a QTc-prolonging drug (e.g., hypocalcemia, hypokalemia, hypomagnesemia)
* History of severe hypersensitivity reaction (≥ grade 3) to any component of the investigational drugs or excipients
* Unable to undergo contrast-enhanced MRI
* Patients who have been treated with any investigational agent(s) within 28 days of the first day of administration of study drugs
* Current active second malignancy other than non-melanoma skin cancers and post-treatment of localized prostate cancer. Patients are not considered to have a currently active malignancy if they are in complete remission for > 3 years prior to study
* Known HIV infection, active Hepatitis B or C infection
* Any ongoing toxicity from prior anti-cancer therapy that is > grade 1 and/or that is progressing in severity (except alopecia) and delayed recovery following last temozolomide cycle
* Additional anti-cancer treatment for glioblastoma other than study drug and supportive measures (i.e. dexamethasone)
* Patients refusing consent for registration, storage, and processing of individual disease characteristics, information on the course of the disease, and information obtained from the family physician and/or other physicians involved in the treatment of the patient about study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Endpoint for phase Ib is the number of patients experiencing dose-limiting toxicity defined as: | Week 12
  * either any unmanageable grade 3-4 toxicity at the end of the second treatment cycle
  * or inability to receive at least 7 of the 10 drugs, all of them being given at ≥50% of the target doses at the end of the second treatment cycle
  * Modifications in terms of doses and/or number of drugs are accepted at any time during treatment.
Endpoint for phase IIa of the trial is objective stable disease or a better tumor response (i.e., partial response, complete response) | Week 12
  as assessed by non-contrast and contrast-enhanced standard cranial MRI interpreted using RANO criteria after 6 treatment cycles in comparison to the baseline MRI.

SECONDARY OUTCOMES:
Overall survival according to Kaplan-Meier estimates | through study completion, an average of 1 year
Progression-free survival according to Kaplan-Meier estimates | through study completion, an average of 1 year
Best tumor response according to the Revised Assessment in Neuro-Oncology (RANO) criteria | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Eric Halatsch, MD, Principal Investigator — Universitiy of Ulm School of Medicine
Locations (1):
- University of Ulm School of Medicine, Ulm, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Halatsch ME, Dwucet A, Schmidt CJ, Muhlnickel J, Heiland T, Zeiler K, Siegelin MD, Kast RE, Karpel-Massler G. In Vitro and Clinical Compassionate Use Experiences with the Drug-Repurposing Approach CUSP9v3 in Glioblastoma. Pharmaceuticals (Basel). 2021 Nov 29;14(12):1241. doi: 10.3390/ph14121241. PMID 34959641
- [Derived] Romo-Perez A, Dominguez-Gomez G, Chavez-Blanco A, Taja-Chayeb L, Gonzalez-Fierro A, Garcia-Martinez E, Correa-Basurto J, Duenas-Gonzalez A. BAPST. A Combo of Common Use Drugs as Metabolic Therapy for Cancer: A Theoretical Proposal. Curr Mol Pharmacol. 2022;15(6):815-831. doi: 10.2174/1874467214666211006123728. PMID 34620071